CLINICAL TRIAL: NCT02433847
Title: Effect of Mosapride on Gut Transit in Patients With Chronic Constipation or Constipated Irritable Bowel Syndrome and Healthy Subjects
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mosa_GIFx_1.0
Record Dates: First submitted 2015-04-13; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Constipated Irritable Bowel Syndrome; Chronic Constipation; Healthy
Keywords: mosapride
MeSH Terms: interventions — mosapride

ARMS (1):
- mosapride (Experimental)
  Interventions: Drug: Mosapride

INTERVENTIONS:
Drug: Mosapride

SUMMARY:
Effect of mosapride 30mg/day on the small bowel and colon transit time in patients with chronic constipation or constipated irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Functional constipation or constipated irritable bowel syndrome patients according to Rome III criteria

Exclusion Criteria:

* Intolerable or hypersensitive to mosapride
* Known Parkinson's ds
* Cardio- or cerebrovascular disease within 3 months
* Malignancy requiring surgery or chemotherapy or radiation within 5 years
* History of GI surgeries except hernia repair, appendectomy, primary closure due to perforation
* Refractory diabetes mellitus/hypertension/thyroid diseases
* Symptomatic heart failure, renal failure, arrhythmia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
colonic transit time | 2 weeks
  the change of colonic transit time after mosapride 30mg/day administration
  : whole colonic transit time, rt. colon / lt. colon / rectosigmoid colonic transit time